CLINICAL TRIAL: NCT01678027
Title: Helicobacter Pylori Eradication to Prevent Gastric Cancer in Subjects With Family History of Gastric Cancer: A Randomized Controlled Study
Brief Title: Gastric Cancer Prevention in the Family Members by Helicobacter Pylori Eradication
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Il Ju Choi, M.D., Ph.D, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NCCCTS04-103
Record Dates: First submitted 2012-08-17; First posted 2012-09-03 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer; Helicobacter Pylori Infection; Family Members
Keywords: Stomach neoplasm; Helicobacter pylori
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo for LAC triple therapy
  Interventions: Drug: Placebo
- LAC triple therapy (Active Comparator): PPI (Lansoprazole), Clarithromycin, Amoxicilline
  Interventions: Drug: LAC triple therapy

INTERVENTIONS:
Drug: Placebo — Lansoprazole placebo, amoxicillin placebo, and clarithromycin placebo, all twice a day for 1 week.
  Arms: Placebo
Drug: LAC triple therapy — Lansoprazole 30 mg, amoxicillin 1,000 mg, and clarithromycin 500 mg, all twice a day for 1 week.
  Other Names: PPI-Clarithromycin containing triple therapy
  Arms: LAC triple therapy

SUMMARY:
This study evaluate whether treatment of Helicobacter pylori infection reduces the incidence of gastric cancer in subjects with family history of gastric cancer.

DETAILED DESCRIPTION:
Helicobacter pylori infection is associated with gastric cancer in epidemiological studies. However, it is still unknown whether H. pylori eradication is useful and required to prevent gastric cancer.

Gastric cancer risk is increased in family members of gastric cancer patient. Though there is no direct evidence that H. pylori infection is a risk factor for gastric cancer in family members of gastric cancer, current European guideline recommends H. pylori eradication in first-degree relatives of gastric cancer patients.

In this study, the investigators will evaluate whether H. pylori eradication can reduce gastric cancer risk in the first-degree family members of gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Sibling or offspring of patients with gastric adenocarcinoma confirmed by EGD and biopsy
* Informed consent should be signed

Exclusion Criteria:

* Gastric cancer history
* Other malignancy within the past 5 years
* Hereditary cancer family member (HNPCC, FAP)
* Peptic ulcer history
* Peptic ulcer, esophageal cancer, gastric cancer case found at EGD
* H. pylori eradication treatment history
* Previous serious side effect to antibiotics
* Serious concurrent infection or nonmalignant disease such as liver cirrhosis, renal failure, cardiovascular diseases
* Pregnant or nursing women
* Psychiatric disorder that would preclude compliance, alcoholics
* Refuse informed consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1838 (Actual)
Dates: Start 2004-11; Primary Completion 2018-12 (Actual); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Gastric cancer incidence | 6 years after last participant enrollment
  The incidence of gastric cancer will be compared between the two arms as the participant assigned into either LAC treatment group or placebo group regardless the final H. pylori infection status.
  Currently, efficacy of LAC triple therapy shows about 75-85% eradication rate of the H. pylori.

SECONDARY OUTCOMES:
Gastric dysplasia incidence | 6 year after last participant enrollment
  Incidence of gastric dysplasia according to the H. pylori treatment
Gastric cancer incidence between H. pylori treatment and H. pylori uninfected groups | 6 year after last participant enrollment
  Gastric cancer incidence between H. pylori treatment group and H. pylori uninfected group
Gastric cancer incidence according to H. pylori status | 6 year after last participant enrollment
  Gastric cancer incidence between H. pylori eradicated group and H. pylori persistent group
All-cause mortality | 6 year after last participant enrollment
  All-cause mortality between H. pylori treatment group and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Il Ju Choi, M.D., Ph.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi IJ, Kim CG, Lee JY, Kim YI, Kook MC, Park B, Joo J. Family History of Gastric Cancer and Helicobacter pylori Treatment. N Engl J Med. 2020 Jan 30;382(5):427-436. doi: 10.1056/NEJMoa1909666. PMID 31995688